CLINICAL TRIAL: NCT01968005
Title: A Randomized, Multi-Center, Double-Blind, Placebo-Controlled Phase III Trial to Evaluate the Efficacy, Tolerability and Safety of Etoreat®(Etodolac-Lidocaine Topical Patch) in the Treatment of Acute Low Back Pain
Brief Title: Etodolac-Lidocaine Patch in the Treatment of Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDRx USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRX-7EAT-1009
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Therapy with placebo
  Interventions: Drug: Placebo
- Etoreat®(Etodolac-Lidocaine Topical Patch) (Experimental): Therapy with experimental drug
  Interventions: Drug: Etoreat®(Etodolac-Lidocaine Topical Patch)

INTERVENTIONS:
Drug: Etoreat®(Etodolac-Lidocaine Topical Patch)
  Other Names: Once daily application of Two patches for 14 days
  Arms: Etoreat®(Etodolac-Lidocaine Topical Patch)
Drug: Placebo
  Other Names: Once daily application of Two patches for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy, tolerability and safety of Etoreat®(Etodolac-Lidocaine Topical Patch) in the treatment of acute low back pain (LBP).

ELIGIBILITY:
Inclusion Criteria:

* Females of child bearing potential must have a negative pregnancy test and be using an adequate method of birth control.
* Subject has an exacerbation of acute low back pain with the onset of the current episode ≥3 and ≤7 days preceding the screening visit. The acute back pain must be muscular in origin.
* Subject has a Current Pain Intensity

Exclusion Criteria:

* Subjects with LBP potentially associated with a specific spinal cause (e.g. known high-grade spondylolisthesis [Grade 3 or 4], tumour, infection, vertebral compression fracture [history ≤1 year], Paget's disease, osteoporosis, spinal stenosis).
* Any past low-back surgery, or scheduled low back surgery during the trial, or any other scheduled surgery or painful procedure during the course of the trial that, in the opinion of the investigator, may affect efficacy or safety assessments.
* Invasive procedures (e.g. epidural injections, spinal cord stimulation therapy) within the past six months aimed to reduce LBP.
* Clinically relevant history of hypersensitivity, allergy or contraindications to any of the IPs' excipients, or to aspirin-like drugs
* Presence of conditions other than LBP that in the investigator's opinion could confound the assessment or self-evaluation of pain, such as but not limited to anatomical deformities, significant skin conditions such as infections (abscesses or ulcers), unilateral or bilateral lower limb pain independent from the indication LBP, painful venous insufficiency, painful post thrombotic syndrome, painful osteoarthritis of the knee, distal lower limb inflammation, or diffuse widespread pain such as fibromyalgia.
* Subject has received passive physical therapy treatments (e.g. deep heat or ultrasound) or used iontophoresis for the pain within the past 12 hours; or requires continued use of an immobilization device for treatment of the current episode of low back pain. Subject on any therapeutic exercise regimen should stay on the same regimen for the duration of the study.
* Subject has used oral pharmacologic treatment (NSAIDs or analgesic medications) less than 5 half-lives before the baseline assessments; acetaminophen or ibuprofen is permitted prior to baseline as long as it is not within six hours of the baseline assessment. Aspirin (81-325 mg daily) taken prophylactically for cardiovascular reasons is permitted.
* Subject has used any form of opioid within 24 hours of study entry or use of opioids for five or more consecutive days within the 30 days preceding enrolment.
* Subject has received systemic corticosteroids in the 30 days preceding the screening visit (e.g. oral, or parenteral administration) or local injections such as intra-articular, peri-tendinous (topical acceptable, unless applied to the target effected area and inhaled or intranasal steroids acceptable, e.g. Flonase®)
* Subject has recently initiated sleep medications, muscle relaxants, anticonvulsants or antidepressants (within the past 30 days); if using any of these, subject must be on a stable dose and regimen for 30 days prior to study enrolment.
* Subject has used TNF-alpha blockers of any type or Class 1 anti-arrhythmic drugs within the past 60 days.
* Subject has a history or physical assessment finding of clinically significant GI ulcers or abnormal bleeding, anemia, kidney disease, liver disease, poorly controlled lung, stomach, heart or other vital organ disease as determined by the study investigator/physician.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
SPID (Summed pain intensity difference) from baseline over the pain assessments from Day 1 to Day 8 | 8 days

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Carlsbad, California
  - Miami, Florida
  - New York, New York
  - Zanesville, Ohio
  - Dallas, Texas
  - El Paso, Texas
  - San Antonio, Texas